CLINICAL TRIAL: NCT03025646
Title: Feasibility of Implementing a Mental Health Care Program and Home-based Training for Mothers of Children With Autism Spectrum Disorder in an Urban Population in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); National Institute of Mental Health (NIMH) (NIH); National Institute of Neurosciences Hospital (NINS) (Other); Institute of Paediatric Neurodisorder and Autism (IPNA) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-16070
Record Dates: First submitted 2017-01-02; First posted 2017-01-19 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-02

CONDITIONS: Maternal Depression
Keywords: Maternal depression; ASD; Home based training program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mental Health care services & home based training — From day 0 of the study period we will initiate setting up the intervention in two schools, which will include two components:
  1. Implementing mental health care services at schools targeting the mothers diagnosed as having depression who have consented to participate in the study (intervention mother).
     Psychologists will provide counseling session over 4-6 months period. Every month a psychiatrist will visit each school for reviewing the records of the mothers and mothers will be referred to the National Institute of Mental Health (NIMH) if necessary
  2. Organizing training sessions of the intervention mothers for supporting enhanced child care at home.
  Organizing training of the intervention mothers by special educator through a parental training module in the schools. Special educator will conduct refresher training at home every month.
  Other Names: psycho social management; home based training program

SUMMARY:
Background (brief):

The global burden of depression accounts for 2.5% of global DALYs, and in South Asia the estimate is 13.3 % of DALYs per 100,000 populations. Mothers of children with Autism Spectrum Disorder (ASD) have reported higher level of depression than mothers of children with other developmental disorder and the prevalence of ASD is high in Asian countries. In Bangladesh 16% of adults suffer from depression and a recent study conducted in Bangladesh has documented a high prevalence of depression among mothers of children with ASD (45%). Mothers are the life time care givers of children with ASD, and a high burden of depression is likely negatively impact on the ability of the mothers to provide care to children at home. Mental health is not addressed in Bangladesh and there is scarcity of qualified providers.

Objectives:

The investigators propose to pilot the feasibility of a package intervention including implementation of mental health care and home based training program for the mothers of children with ASD integrated in the regular activities of the special schools that offer ASD care in Dhaka city in Bangladesh.

Methods:

The study will be conducted in 2 selected special schools over 15 months. In the first stage, the investigators will set up the study in two schools and identify various stakeholders for qualitative assessment of the barriers of implementing the intervention at the institutional level, individual level, family level, provider level, policy maker level and at the level of the state. Research staff will identify mothers 18 years of age or older who has a child with ASD between 3 and 17 years of age enrolled in the school. Following consent, data collector will obtain data and assess current major depressive episode (MDE) of the eligible mothers following a standard diagnostic tool (SCID-I). All mothers diagnosed as having MDE will be invited to participate in the intervention (intervention mothers) and the investigators will assess the performances in children with ASD by applying ASD Diagnostic Check-list (ADCL).

In the second stage, investigators will implement interventions over 4-6 months, including (a) implementing mental health care services at the selected schools targeting the intervention mothers, and (b) organizing training sessions of the intervention mothers for supporting child care at home for enhancing child performances. Every month a psychiatrist will visit each school for providing necessary advice and treatment to the intervention mothers or suggest referral to hospital care, if necessary.

One special educator will be deployed at each school who will organize structured training sessions for educating the intervention mothers by using BCC materials developed and validated by icddr,b in the local setting. The special educators will conduct multiple group sessions including 5-8 mothers in each group for covering the 6 modules over 2 weeks time, and follow up intervention mothers at home every month for conducting refresher's training, documenting the need of additional training supports, and linking mother with an ASD expert for helping mothers taking a decision.

In stage 3, investigators will conduct post intervention qualitative survey with various stakeholders who would be involved with implementing the intervention and participated in the baseline qualitative survey. End line assessment will be conducted of current major depressive episode (MDE) among all mothers and assess the performance of the children of intervention mothers in order to assess the impact of the training at home.

Outcome measures/variables:

The primary outcome of the study is to assess the feasibility of institutionalizing the combined intervention of mental health care supports and the home based training program of the mothers who would be diagnosed as having major current major depressive episode. The primary outcome will be assessed by obtaining the perspectives of various stakeholders. The following parameters will be assessed for measuring feasibility of the proposed intervention.

Acceptability, Adaptability, Demands, Practicality, Implementation, Integration

The secondary outcomes will include estimating the impact of the combined interventions on the prevalence rate of maternal depression (MDE), individual performances of children, and cost of intervention. Adaptation of the proposed strategy, if feasible will help the mothers of children with ASD become skilled workforces for filling in the gap of the special educators in resource poor settings, and extension of these services to more children with ASD.

DETAILED DESCRIPTION:
The study will be conducted in 2 selected special schools in Dhaka city, (i) Autiam welfare Foundation (AWF: http://awfbd.com/) and (ii) Society for the Welfare of Autistic Children (SWAC: http://www.ASDbd.com/swac-bd/) who have more than 10 years of experiences with offering quality services for ASD care in Bangladesh. The investigator will conduct the study in both schools in 3 stages:

* Preparatory phase and baseline assessment (stage 1)
* Implementation of intervention (stage 2)
* End line assessment (stage 3)

Stage 1:

The investigator will set up the study in two schools and identify various stakeholders including the managers of the schools, special educators, psychologists, psychiatrists, medical doctors, parent of children with ASD, policy makers etc. Data collector will obtain written const from them and conduct in depth interviews for assessing barriers of implementing the intervention at institutional level, individual level, family level, provider level, policy makers level and at the level of the state prior to intervention.

Research staff will identify those mothers who are at least 18 years of age and has a child with ASD between 3 and 17 years of age enrolled in the school. The staff in the intervention phase would not be involved in the baseline or end line surveys. The investigator will recruit separate staff for conducting baseline and end line surveys. Data collector will obtain additional school based information regarding the children's ASD diagnosis and an expert from IPNA will reconfirm their ASD by ADCL in order to further validate and rate the ASD diagnoses with health and education related information.

Data collector will obtain written consent from the eligible mothers who have child with ASD and obtain essential socio demographic and other relevant data, and perform clinical diagnosis of major depressive disorder (MDD) and current major depressive episode (MDE) following a standard diagnostic tool (SCID-I) based on DSM-IV criteria as it has already been validated through several studies in Bangladesh. All mothers diagnosed as having MDE will be invited to participate in the intervention following a written consent (intervention mothers). However, any mother identified with severe forms of depression with any suicidal ideation or unsafe thoughts will be referred for urgent hospital based mental health services in the community (as per standard of care and ethical obligations), and they will not be invited to participate in the study. The selected schools would have at least 100-150 children with ASD enrolled in a given year, and we anticipate that a total of ~ 54 to 80 mothers will participate in the intervention. Data collector will interview the intervention mothers in order to assess the individual performances of their children by using a standard tool ADCL (ASD Diagnostic Check-list). ADCL is a standard tool applied by ASD experts in Bangladesh to track improvement in performances in children with ASD [22].This tool comprises of 60 items focusing on 6 major areas of ASD, including (i) General Observation (13 items), (ii) Cognition (10 items), (iii) Emotion (8 items), (iv) Social/Self Help (8 items), (v) Communication (12 items), and (vi) Sensory deficiency (9 items).

Stage 2:

From day 0 of the study period investigator will initiate setting up the intervention in two schools, which will include two components; (a) Implementing mental health care services at schools targeting the mothers diagnosed as having depression who have consented to participate in the study (intervention mother) and (b) Organizing training sessions of the intervention mothers for supporting enhanced child care at home. Although the mental health services will target mothers who would volunteer to participate in the intervention. The proposed intervention will be implemented over 4-6 months period; the two components of the package have been described below in details.

1. . Implementing mental health care services at school

   The investigator will develop a counseling centre at each school by deploying one trained female psychologists who would provide counseling to the intervention mothers. Investigator will adopt the psychological management procedures that have been commonly administered by the experts of National Institute of Mental Health, Bangladesh (NIMH, B). Intervention guidelines will be submitted to ERC for reviewing and necessary approval of the document before the final application in the study. The mental health services counseling module will comprises of the following topics:
   1. Psycho education

      Psycho education refers to the education offered to individuals with a mental health condition and their families to help empower them and deal with their condition in an optimal way. Psycho education will be given by a trained psychologists under the guidance of a psychiatrists to increase the self esteem of the mothers, which will include the brief concept on depression, the probable etiology, how to mitigate the symptoms, compliance to the therapeutic process and the consequences. This method of psychological management is commonly practiced by the psychologists and also has been used in the former studies in Bangladesh.
   2. Assessment of the strength and weakness of the mothers

      The psychologists will assess the strengths and weakness of the mothers, and discover their personal obstacles, issues that might hinder their progress in terms of social context, family support, financial state, educational qualification, empowerment etc.
   3. Sharing the management plan with the mothers The psychologists will share the whole management processes with the mothers and any opinion from the mother could be a part of the management. The goal is to empower mothers and include them as a part of the management team counseling other mothers.
   4. Reconstruction of the cognition Cognitive restructuring is a psychotherapeutic process of learning to identify and dispute irrational or maladaptive thoughts known as cognitive distortions. It is a core part of Cognitive Behavioral Therapy (CBT). CBT is a structured method and one of the most effective psychological treatments commonly used by the psychiatrists and psychologists of Bangladesh to intervene depression. To manage depression minimum 12 sessions are required which can be more upon the severity of the clients. CBT mainly deals with exploring problems, thoughts, feelings and behavior of the clients. It is one of the major components of our intervention protocol based on the standard practice of the experts of Bangladesh.
   5. Behavior therapy- graded activity Graded activity is a principle of therapeutic intervention in which tasks are classified and gradually presented according to the client's level of function and the challenge or degree of skill (physical, social, or cognitive) required by the task. In this study after assessing the strengths and weaknesses of the mothers their functional activity also be monitored and will try to increase. The graded activity starts from personal care, daily household activities, child care, engagement in small and easy tasks and complex and productive tasks.
   6. Developing a mother's community and engaging depressed mothers in community related activities

   The psychologist will arrange a workshop in each participating school at two months interval for enabling mothers meet other mothers in the intervention and create a common platform where they can share their experiences , success stories and encourage a positive reinforcement on the depressed mothers. The mothers will be encouraged to participate in the social awareness or other activities arrange by the schools, so that the mothers refrain from social isolation and rebuild their self esteem.

   Every month a psychiatrist of NIMH, B will visit each school for reviewing the records maintained by the psychologist and provide necessary advice to the psychologist for additional care of the depressed mother as and when required. The psychiatrist will reassess the additional need of a mother following face to face consultation if suggested by the record review, or identified by the psychologist. The medical care will specially focus on management of depression with varying degree of severity as listed below, including care for common mental disorders (neurosis), if exists. Mothers will be referred to the National Institute of Mental Health for providing advanced mental health care if necessary and be provided with free medicines that are available at the NIMH including anti- depressant, anxio-lytic, anti-psychotic etc.

   The medical care will follow the management guideline adopted in NIMH for treating the following conditions, including referral to the National Institute of Mental Health for advanced mental health care if necessary.

   If mild to moderate: field psychologist: counseling and Cognitive behavior therapy.

   If moderate to severe (without suicidal tendency): Counseling and Cognitive behavior therapy. Drugs prescribed by psychiatrists during the periodical visits at the school. If mothers have a suicidal tendency she will be immediately referred to NIMH or other collaborative institutes. For other psychiatric disorders, such as, major mental disorder or psychosis), the psychiatrist will prescribe drugs during their periodic visits and refer a mother to NIMH or any other hospital that a mothers prefers, if fund necessary by the discretion of the psychiatrist.
2. Organizing training of the intervention mothers in the schools for supporting child care at home A parental training module was developed in the local language (Bangla) by icddr,b led by Naheed et al in 2015 and customized according to the local context under the guidance of an Expert Working Group comprised of experts in various relevant disciplines. The module was piloted with 56 parents and validated for its application in the local setting. Investigator will deploy one special educator at each school who will organize structured training sessions for the intervention mothers by using BCC materials. The special educator will conduct multiple group sessions including 5-8 mothers in each group for covering the 6 modules over 2 weeks time. The special educators will follow up with mothers at home every month for conducting refresher's training and document the need of additional training supports for an individual child as advised by the mother or observed by the educator herself. The special educator will consult with one of the Co Investigators who is an ASD expert and incorporate necessary aids or additional training for a specific child as advised by the expert, and link mother with the ASD expert for helping mothers taking a decision.

Estimating the cost of the pilot intervention

The project will estimate the overall costs that would incur to an individual institution due to introduction of the combined services at the school. As such, research staff will track costs of mental health services throughout the intervention period of 6 months and cost of conducting training of mothers at school over 4 months period. Costs related to mental health services will include counseling sessions, psychiatrists' visits, facility, training, special educators, training materials and any other cost that might be potentially borne by the institutions.

Stage 3:

This will also include a qualitative end line survey conducted with the intervention mothers, special educators, psychologists, psychiatrists and principals of the school who would be involved with implementing the intervention and participated in the baseline qualitative survey. The end line qualitative survey will assess views of various stakeholders about the directions for institutionalizing the proposed intervention based on their experiences in the intervention, particularly aligned with the barriers documented during the intervention period. Research staff will also conduct an end assessment of current major depressive episode (MDE) among all mothers in the selected schools including the mothers participated in the intervention, and assess the performance level and degree of ASD in their children to assess the impact of the training module.

Survey for the maternal depression

Inclusion criteria:

1. Managers, special educators, psychologists, therapists, depressed mothers, and family members of the depressed mothers
2. Psychiatrists, Pediatricians, medical doctors, working in the collaborating medical institutions who are involved with ASD care.
3. Parents of children with ASD enrolled in other schools that offer ASD services.
4. Policy makers who are involved in the Ministry of Health, the Ministry of Family Welfare, Autism cell etc. for developing the national strategic plan and policies for strengthening ASD care in Bangladesh. .

Exclusion Criteria:

1. Participants who are too ill to commute
2. Participants who are mentally compromised to give a voluntary consent for her own.

Research staff will conduct in depth interviews with the above listed participants for assessing barriers of implementing the intervention at institutional level, individual level, family level, provider level, policy makers level and at the level of the state prior to intervention.

Intervention Phase:

Inclusion criteria:

Psychologists will identify those mothers who would be diagnosed as having a current major depressive episode (MDE) at the baseline survey as assessed by PHQ-9 and SCID, and willing to participate in the intervention for the next 6 months.

Exclusion Criteria:

Any mother diagnosed as having a severe forms of depression with any suicidal ideation or unsafe thoughts will be referred for urgent hospital based mental health services in the community (as per standard of care and ethical obligations), and will not be invited to participate in the study or will be withdrawn from the study if such a condition develops in the course of intervention.

ELIGIBILITY:
Inclusion Criteria:

Survey for the maternal depression

Inclusion criteria:

1. Managers, special educators, psychologists, therapists, depressed mothers, and family members of the depressed mothers
2. Psychiatrists, Pediatricians, medical doctors, working in the collaborating medical institutions who are involved with ASD care.
3. Parents of children with ASD enrolled in other schools that offer ASD services.
4. Policy makers who are involved in the Ministry of Health, the Ministry of Family Welfare, Autism cell etc. for developing the national strategic plan and policies for strengthening ASD care in Bangladesh.

Intervention Phase:

Inclusion criteria:

We will identify those mothers who would be diagnosed as having a current major depressive episode (MDE) at the baseline survey as assessed by PHQ-9 and SCID, and willing to participate in the intervention for the next 6 months.

Exclusion Criteria:

Survey for the maternal depression

1. Participants who are too ill to commute
2. Participants who are mentally compromised to give a voluntary consent for her own.

Intervention Phase:

Any mother diagnosed as having a severe forms of depression with any suicidal ideation or unsafe thoughts will be referred for urgent hospital based mental health services in the community (as per standard of care and ethical obligations), and will not be invited to participate in the study or will be withdrawn from the study if such a condition develops in the course of intervention.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Participants who can accept, afford and adapt the implemented program of mental health service and home based training program | 6 months
  assessed by qualitative guideline thorough IDI, KII

SECONDARY OUTCOMES:
Number of mothers with Major Depressive Disorder (MDD) | 6 months
  assessed by SCID-I
Number of children with ASD who have improved their skill in terms of communication, behavior and social skills | 6 months
  assessed by ADCL (ASD Diagnostic Check-list)

CONTACTS AND LOCATIONS:
Locations (1):
- Awf, Swac, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No